CLINICAL TRIAL: NCT00716885
Title: The Effect of Left Ventricular Filling Pressure on Pulmonary Clearance of Free Radical Loaded White Blood Cells and Platelets in Congestive Heart Failure Patients Before and After Biventricular Pacing
Acronym: OXIS-PACING
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Professor dr. Walter J. Paulus, VU University Medical Center
Other Study IDs: 1781
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-05

CONDITIONS: Congestive Heart Failure
Keywords: Heart failure; Oxidative stress; Endothelial Progenitor Cells; White blood cells
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloodsamples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CHF: Informed consented participants are recruited among all patients admitted to the OLVG hospital.
  Inclusion criteria:
  * Chronic congestive heart failure patients of all ages selected for biventricular pacemaker implantation for resynchronization therapy
  * Dyspnoe NYHA class III and IV
  * Optimal and constant heart failure treatment according to the ESC guidelines
  Exclusion criteria:
  * Renal failure (creatinine >1.70 mg/dl)
  * Signs of infection or inflammation
- Control: The control group consists of ten age-matched volunteers with a normal left ventricular ejection fraction and without signs or symptoms of heart failure.

SUMMARY:
1. To assess whether a correlation exist between the degree of pulmonary clearance of free radical positive white bloodcells and platelets and the degree of pulmonary congestion in congestive heart failure (CHF) patients
2. To asses whether cardiac resynchronization therapy improves pulmonary clearance of free radical positive white blood cells and platelets in CHF patients by alleviating pulmonary congestion
3. Interaction of oxidative stress with circulating endothelial progenitor cells (EPCs) and presence of apoptotic endothelial (progenitor) cells

DETAILED DESCRIPTION:
Evidence exists that oxidative stress is enhanced in congestive heart failure patients resulting in damage to cellular lipids, proteins and DNA. Because of free radical-induced apoptosis of skeletal muscle fibers, oxidative stress is an important contributor to skeletal muscle fatigue and low exercise tolerance of congestive heart failure patients. Enhanced oxidative stress in congestive heart failure can exert negative inotropic effects and can have important effects on the structure and function of the myocardium, and may be implicated in the progression of congestive heart failure. Free radical stress could also impair recruitment and differentiation of circulating endothelial progenitor cells resulting in increased all cause mortality.

Reduced pulmonary clearance of free radical loaded white blood cells and platelets is an important contributor to enhanced oxidative stress in congestive heart failure patients. Failure of pulmonary clearance of free radical loaded white blood cells and platelets probably results from pulmonary congestion which has led to the rationale of the current study. Biventricular pacing for resynchronization therapy in congestive heart failure patients reduces left ventricular filling pressure and pulmonary congestion. Biventricular pacing may therefore augment pulmonary clearance of free radical loaded white blood cells and platelets in congestive heart failure patients.

We conduct a prospective, observational clinical study to investigate the correlation of left ventricular filling pressure, pulmonary clearance of FR loaded circulating white blood cells and platelets and number of endothelial progenitor cells in congestive heart failure (CHF) patients before and after implantation of a biventricular pacemaker for resynchronization therapy.

ELIGIBILITY:
Patient selection

Informed consented participants are recruited among all patients admitted to the OLVG hospital.

Inclusion criteria:

* Chronic congestive heart failure patients of all ages selected for biventricular pacemaker implantation for resynchronization therapy
* Dyspnoe NYHA class III and IV
* Optimal and constant heart failure treatment according to the ESC guidelines

Exclusion criteria:

* Renal failure (creatinine > 1.70 mg/dl)
* Signs of infection or inflammation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the OLVG hospital for worsening congestive heart failure selected for biventricular pacemaker implantation
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
• Number of (apoptotic) endothelial (progenitor) cells | baseline

SECONDARY OUTCOMES:
• Oxidative stress: cytosolic and mitochondrial FR | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- OLVG Hospital, Amsterdam, North Holland, Netherlands

REFERENCES:
- See also: United Committee Human Research (the Netherlands) — http://www.vcmo.nl